CLINICAL TRIAL: NCT02260362
Title: Observatory of Pulmonary Arterial Hypertension of Congenital Heart Disease
Acronym: ItinerAir
Status: Completed | Type: Observational
Sponsor: French Cardiology Society (Other)
Responsible Party: Sponsor
Other Study IDs: 14126
Record Dates: First submitted 2014-10-06; First posted 2014-10-09 (Estimated); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Pulmonary Arterial Hypertension of Congenital Heart Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HTAP of Congenital Heart Disease

SUMMARY:
The complex congenital cardiac malformations are a significant number of different diseases, each having specific natural histories. The interface with pulmonary arterial hypertension (HTAP) is high since the physiology of many of these disorders comprises alterations in pulmonary vasculature.

This observatory is a cohort of 400 patients enrolled in 3 years, older than one month, having been informed and have agreed to participate in the study and with congenital heart disease other than patent foramen ovale as well as a diagnosis of pulmonary hypertension confirmed by cardiac catheterization.

The main objectives of this report are to know

* Incidence of congenital heart disease in HTAP France.
* Describe the natural history of HTAP in a large population of patients Congenital heart disease in France
* The characteristics of HTAP congenital heart disease
* Having a cohort study

ELIGIBILITY:
Inclusion Criteria:

* The patient has a congenital heart disease other than patent foramen ovale
* The diagnosis of pulmonary hypertension was confirmed by cardiac catheterization. Only patients with Eisenmenger syndrome can be included without catheterization.
* The catheterization was done after 1 January 2009
* A mean pulmonary artery pressure > 25 mm Hg
* Pulmonary vascular resistances > 3 piece Wood m2
* Pulmonary capillary pressure available
* Consent for inclusion in the study must be signed by parents or legal guardians for minors, by the patient for adults.
* The patient he had a surgical procedure or interventional catheterization cardiac catheterization between his diagnosis and inclusion in the observatory? If yes, it can only be included if a new catheterization confirmed the persistence of HTAP at least 6 months after the procedure.
* Patient follow-up (at least once a year) in the center for its HTAP associated with congenital heart disease its

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with Pulmonary Arterial Hypertension of Congenital Heart Disease supported by one of the 20 centers participating in the observatory during the period incusion and respecting al the selection criteria
Sampling Method: Non-Probability Sample
Enrollment: 349 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Incidence HTAP of congenital heart disease in France. | 3 years
  Number of HTAP of congenital heart disease in France after 3 years of inclusions

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Necker Enfants Malades, Paris, France

REFERENCES:
- [Background] Berger RM, Beghetti M, Humpl T, Raskob GE, Ivy DD, Jing ZC, Bonnet D, Schulze-Neick I, Barst RJ. Clinical features of paediatric pulmonary hypertension: a registry study. Lancet. 2012 Feb 11;379(9815):537-46. doi: 10.1016/S0140-6736(11)61621-8. Epub 2012 Jan 11. PMID 22240409
- [Background] Barst RJ, McGoon MD, Elliott CG, Foreman AJ, Miller DP, Ivy DD. Survival in childhood pulmonary arterial hypertension: insights from the registry to evaluate early and long-term pulmonary arterial hypertension disease management. Circulation. 2012 Jan 3;125(1):113-22. doi: 10.1161/CIRCULATIONAHA.111.026591. Epub 2011 Nov 15. PMID 22086881
- [Background] Barst RJ, Ivy DD, Foreman AJ, McGoon MD, Rosenzweig EB. Four- and seven-year outcomes of patients with congenital heart disease-associated pulmonary arterial hypertension (from the REVEAL Registry). Am J Cardiol. 2014 Jan 1;113(1):147-55. doi: 10.1016/j.amjcard.2013.09.032. Epub 2013 Oct 4. PMID 24176071
- [Background] Humbert M, Sitbon O, Chaouat A, Bertocchi M, Habib G, Gressin V, Yaici A, Weitzenblum E, Cordier JF, Chabot F, Dromer C, Pison C, Reynaud-Gaubert M, Haloun A, Laurent M, Hachulla E, Simonneau G. Pulmonary arterial hypertension in France: results from a national registry. Am J Respir Crit Care Med. 2006 May 1;173(9):1023-30. doi: 10.1164/rccm.200510-1668OC. Epub 2006 Feb 2. PMID 16456139
- [Background] Fraisse A, Jais X, Schleich JM, di Filippo S, Maragnes P, Beghetti M, Gressin V, Voisin M, Dauphin C, Clerson P, Godart F, Bonnet D. Characteristics and prospective 2-year follow-up of children with pulmonary arterial hypertension in France. Arch Cardiovasc Dis. 2010 Feb;103(2):66-74. doi: 10.1016/j.acvd.2009.12.001. Epub 2010 Feb 11. PMID 20226425
- [Background] van Loon RL, Roofthooft MT, Hillege HL, ten Harkel AD, van Osch-Gevers M, Delhaas T, Kapusta L, Strengers JL, Rammeloo L, Clur SA, Mulder BJ, Berger RM. Pediatric pulmonary hypertension in the Netherlands: epidemiology and characterization during the period 1991 to 2005. Circulation. 2011 Oct 18;124(16):1755-64. doi: 10.1161/CIRCULATIONAHA.110.969584. Epub 2011 Sep 26. PMID 21947294
- [Background] Duffels MG, Engelfriet PM, Berger RM, van Loon RL, Hoendermis E, Vriend JW, van der Velde ET, Bresser P, Mulder BJ. Pulmonary arterial hypertension in congenital heart disease: an epidemiologic perspective from a Dutch registry. Int J Cardiol. 2007 Aug 21;120(2):198-204. doi: 10.1016/j.ijcard.2006.09.017. Epub 2006 Dec 19. PMID 17182132